CLINICAL TRIAL: NCT02532283
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Pharmacokinetics, Safety, and Antiviral Activity of JNJ-63623872 in Combination With Oseltamivir in Adult and Elderly Hospitalized Patients With Influenza A Infection
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Antiviral Activity of JNJ-63623872 in Combination With Oseltamivir in Adult, and Elderly Hospitalized Participants With Influenza A Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107746; 2015-003002-17 (EudraCT Number); 63623872FLZ2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Influenza A Virus
Keywords: Influenza A virus; JNJ-63623872; Oseltamivir
MeSH Terms: interventions — pimodivir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-63623872 plus Oseltamivir (Experimental): Participants will be administered JNJ-63623872 600 milligram (mg) tablets and oseltamivir 75 mg capsules orally twice daily for 7 days.
  Interventions: Drug: JNJ-63623872; Drug: Oseltamivir
- Placebo plus Oseltamivir (Experimental): Participants will be administered placebo tablets and oseltamivir 75 mg capsules orally twice daily for 7 days.
  Interventions: Drug: Placebo; Drug: Oseltamivir

INTERVENTIONS:
Drug: JNJ-63623872 — Participants will be administered JNJ-63623872 600 milligram (mg) tablets orally twice daily for 7 days.
  Arms: JNJ-63623872 plus Oseltamivir
Drug: Placebo — Participants will be administered placebo tablets orally twice daily for 7 days.
  Arms: Placebo plus Oseltamivir
Drug: Oseltamivir — Participants will be administered oseltamivir 75 mg capsules orally twice daily for 7 days.

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetic parameters of JNJ-63623872 in combination with oseltamivir in elderly participants (aged 65 to <= 85 years) compared to adults (aged 18 to <= 64 years) with influenza A infection.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled, multicenter (when more than one hospital or medical school team work on a medical research study) study to evaluate the effect of JNJ-63623872 in combination with oseltamivir in participants with influenza A infection. The study consists of 3 Phases: Screening visit (1 Day), participants who meet all eligibility criteria will be randomized in a 2:1 ratio to receive study drug in double-blind treatment Phase (7 Days) and follow up Phase (21 Days). The duration of participation in the study for each participant is approximately 28 Days. Primarily Pharmacokinetic parameters of JNJ-63623872 will be measured. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant requires hospitalization to treat influenza infection and/or to treat complications of influenza infection
* Participant tested positive for influenza A infection within 1 day of signing of the informed consent form (ICF)/assent form using a polymerase chain reaction (PCR)-based rapid molecular diagnostic assay
* Participants must be capable of swallowing study medication tablets and capsules
* Each participant (or their legally acceptable representative) must sign an ICF indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in the protocol

Exclusion Criteria:

* Participant received more than 3 doses of the influenza antiviral medication oseltamivir, zanamivir, or peramivir since the start of the influenza symptoms, or ribavirin within 6 months prior to Screening
* Participant is unwilling to undergo regular nasal Mid-turbinate (MT) swabs or has any physical abnormality which limits the ability to collect regular nasal specimens
* Participant is immunocompromised, whether due to underlying medical condition (example, malignancy) or medical therapy (example, medications, chemotherapy, radiation, post-transplant)
* Participant is undergoing peritoneal dialysis, hemodialysis, or hemofiltration
* Participant has an estimated glomerular filtration rate (eGFR) less than or equal to (<=)30 milliliter (mL)/minute (min)/1.73 meter^2 (m^2) according to the Modification of Diet in Renal Disease (MDRD) equation, assessed at Screening or based on the most recent clinically relevant creatinine value if available

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (68):
- United States (14):
  - Fresno, California
  - Long Beach, California
  - Stanford, California
  - Atlantis, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Teaneck, New Jersey
  - Winston-Salem, North Carolina
  - Houston, Texas
- Australia (3):
  - Cairns
  - South Brisbane
  - Westmead
- Belgium (3):
  - Aalst
  - Brussels
  - Leuven
- Brazil (3):
  - Passo Fundo
  - Porto Alegre
  - São Paulo
- Canada (2):
  - Hamilton, Ontario
  - Québec, Quebec
- France (10):
  - Dijon
  - Grenoble
  - Limoges
  - Lyon
  - Nantes
  - Paris
  - Poitiers
  - Rennes
  - Saint-Priest-en-Jarez
  - Tours
- Germany (2):
  - Donaustauf
  - Jena
- Hong Kong, Hong Kong
- Malaysia (8):
  - Kota Bharu
  - Kuala
  - Kuala Lumpur
  - Kuching
  - Malacca
  - Miri
  - Sungai Buloh
  - Taiping
- Netherlands (3):
  - Rotterdam
  - Utrecht
  - Zutphen
- Hamilton, New Zealand
- Singapore, Singapore
- Spain (9):
  - Alicante
  - Barcelona
  - Bizkaia
  - Elche
  - Granada
  - Madrid
  - Mataró
  - San Sebastián
  - Vigo
- Sweden (3):
  - Malmo
  - Umeå
  - Uppsala
- Turkey (Türkiye) (5):
  - Ankara
  - Eskişehir
  - Istanbul
  - Izmir
  - Trabzon

REFERENCES:
- [Derived] O'Neil B, Ison MG, Hallouin-Bernard MC, Nilsson AC, Torres A, Wilburn JM, van Duijnhoven W, Van Dromme I, Anderson D, Deleu S, Kosoglou T, Vingerhoets J, Rossenu S, Leopold L. A Phase 2 Study of Pimodivir (JNJ-63623872) in Combination With Oseltamivir in Elderly and Nonelderly Adults Hospitalized With Influenza A Infection: OPAL Study. J Infect Dis. 2022 Aug 12;226(1):109-118. doi: 10.1093/infdis/jiaa376. PMID 32604406

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 102 participants were randomized. 3 participants were randomized but not treated due to withdrawal of consent before treatment start. Therefore, the Safety Set, comprising all participants who received at least 1 dose of study drug(s), consisted of 99 participants.
Groups:
- Pimodivir 600 mg Plus Oseltamivir 75 mg: Participants received pimodivir 600 milligram (mg) tablets and oseltamivir 75 mg capsules orally twice daily for 7 days. Dose of oseltamivir was adjusted from 75 mg to 30 mg and vice versa during the course of treatment based on the estimated-glomerular filtration rate (eGFR) value.
- Placebo Plus Oseltamivir 75 mg: Participants received matching placebo tablets and oseltamivir 75 mg capsules orally twice daily for 7 days. Dose of oseltamivir was adjusted from 75 mg to 30 mg and vice versa during the course of treatment based on the eGFR value.
Period: Overall Study
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Started | 64 | 35
Full Analysis Set | 63 | 32
Completed | 55 | 30
Not Completed | 9 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug and analyzed as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg | Total
Number analyzed (Participants) | 64 | 35 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (16.06) | 57.2 (13.71) | 57.8 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 45
  Male | 37 | 17 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 55 | 32 | 87
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 7 | 12
  Black or African American | 6 | 7 | 13
  More than one race | 0 | 1 | 1
  Other | 2 | 1 | 3
  Unknown or Not Reported | 2 | 0 | 2
  White | 48 | 19 | 67
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 3 | 0 | 3
  FRANCE | 6 | 2 | 8
  GERMANY | 0 | 2 | 2
  HONG KONG | 0 | 1 | 1
  MALAYSIA | 3 | 4 | 7
  NETHERLANDS | 3 | 1 | 4
  SINGAPORE | 1 | 0 | 1
  SPAIN | 16 | 7 | 23
  SWEDEN | 8 | 4 | 12
  TURKEY | 6 | 3 | 9
  UNITED STATES | 18 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Pimodivir
Description: Cmax is the maximum observed plasma concentration. As per planned analysis, results are presented by age groups (65 to less than or equal to [<=] 85 years and 18 to <=64 years).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 10 and 12 hours post-dose on Day 3
Population: Pharmacokinetic (PK) analysis set included all participants from whom sufficient concentration data were available to facilitate derivation of at least one PK parameter. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Groups:
- Elderly Adults (65 to Less Than or Equal to [<=] 85 Years); Non-elderly Adults (18 to <=64 Years): Participants received pimodivir 600 mg tablets and oseltamivir 75 mg capsules orally twice daily for 7 days.
Arm/Group | Elderly Adults (65 to Less Than or Equal to [<=] 85 Years) | Non-elderly Adults (18 to <=64 Years)
Number analyzed (Participants) | 15 | 20
Nanogram per milliliter (ng/mL) | 5933 (4427) | 5378 (3888)

2. Primary Outcome: Minimum Observed Plasma Concentration (Cmin) of Pimodivir
Description: Cmin is the minimum observed plasma concentration. As per planned analysis, results are presented by age groups (65 to <= 85 years and 18 to <=64 years).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 10 and 12 hours post-dose on Day 3
Population: PK analysis set included all participants from whom sufficient concentration data were available to facilitate derivation of at least one PK parameter. Here, N (number of participants analyzed) signifies number of participants evaluable for this OM.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Elderly Adults (65 to Less Than or Equal to [<=] 85 Years) | Non-elderly Adults (18 to <=64 Years)
Number analyzed (Participants) | 15 | 21
ng/mL | 738 (892) | 507 (414)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time of Administration to 12 Hours After Dosing (AUC [0-12]) of Pimodivir
Description: AUC (0-12) is the area under the plasma concentration-time curve from time zero to 12 hours after dosing of pimodivir. As per planned analysis, results are presented by age groups (65 to <= 85 years and 18 to <=64 years).
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 10 and 12 hours post-dose on Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*h/mL)
Arm/Group | Elderly Adults (65 to Less Than or Equal to [<=] 85 Years) | Non-elderly Adults (18 to <=64 Years)
Number analyzed (Participants) | 15 | 20
nanogram hours per milliliter (ng*h/mL) | 27386 (25191) | 20101 (11063)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious AEs (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with treatment and therefore can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with use of a medicinal product, whether or not related to that medicinal product. TEAEs were defined as AEs that were reported or worsened on after start of study drug(s) dosing through safety follow-up visit. A serious adverse event (SAE) is any untoward medical occurrence that at any dose resulting in any of following outcomes: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to 28 Days
Population: Safety analysis set included all participants who received at least one dose of study drug(s) and were analyzed by drug received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 64 | 35
Participants
  TEAEs | 48 | 25
  TESAEs | 11 | 4

5. Secondary Outcome: Time to Influenza A Viral Negativity
Description: Time to influenza A viral negativity was determined based on quantitative reverse transcription polymerase chain reaction (qRT-PCR). A participant was considered influenza A viral negative at the time point that the first negative nasal midturbinate (MT) swab was recorded (in days). Viral Load Limit of detection (LOD) = 2.18 log10 viral particles per milliliter (vp/mL). Results less than (<) limit of quantification (LOQ) and greater than (>) LOD (target detected) are imputed with 2.12 log10 vp/mL, results <LOD (target not detected) are imputed with 0 log10 vp/mL.
Time Frame: Up to 14 Days
Population: Full Analysis set (FAS) was defined as all randomly assigned participants who received at least 1 dose of study drug and who had a confirmed infection with influenza A.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 63 | 32
Days | 9.53 [8.55 to 12.68] | 9.74 [6.67 to 12.99]

6. Secondary Outcome: Influenza Viral Load Over Time
Description: Influenza viral load over time (Log 10 viral particles per milliliter [vp/mL]) was measured by qRT-PCR. Viral Load LOD = 2.18 log10 vp/mL. Results < LOQ and > LOD (target detected) are imputed with 2.12 log10 vp/mL and results <LOD (target not detected) are imputed with 0 log10 vp/mL.
Time Frame: Baseline, Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 and 14
Population: FAS was defined as all randomly assigned participants who received at least 1 dose of study drug and who have a confirmed infection with influenza A. Here, N (number of participants analyzed) signifies number of participants evaluable for this OM and 'n' signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Log 10 vp/mL
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 58 | 30
Log 10 vp/mL
  Baseline | 5.45 (1.737) | 5.90 (1.513)
  Day 1: number analyzed (Participants) | 4 | 1
  Day 1 | 6.40 (0.757) | 4.43 (NA) — Here, NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Day 2: number analyzed (Participants) | 57 | 28
  Day 2 | 4.75 (1.290) | 4.63 (1.757)
  Day 3: number analyzed (Participants) | 45 | 24
  Day 3 | 3.83 (1.310) | 3.98 (1.924)
  Day 4: number analyzed (Participants) | 34 | 15
  Day 4 | 3.00 (1.486) | 3.14 (1.806)
  Day 5: number analyzed (Participants) | 55 | 28
  Day 5 | 2.57 (1.716) | 2.60 (1.803)
  Day 6: number analyzed (Participants) | 14 | 6
  Day 6 | 2.07 (1.454) | 2.18 (2.457)
  Day 7: number analyzed (Participants) | 14 | 5
  Day 7 | 1.95 (1.478) | 2.38 (2.212)
  Day 8: number analyzed (Participants) | 55 | 20
  Day 8 | 1.82 (1.709) | 1.43 (1.648)
  Day 9: number analyzed (Participants) | 7 | 1
  Day 9 | 1.51 (1.034) | 0.00 (NA) — Here, NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Day 10: number analyzed (Participants) | 54 | 23
  Day 10 | 1.39 (1.676) | 0.99 (1.295)
  Day 11: number analyzed (Participants) | 6 | 1
  Day 11 | 0.42 (1.017) | 0.00 (NA) — Here, NA indicates that data was not available as standard deviation could not be calculated for a single participant.
  Day 12: number analyzed (Participants) | 2 | 0
  Day 12 | 1.06 (1.499) |
  Day 13: number analyzed (Participants) | 2 | 0
  Day 13 | 1.06 (1.499) |
  Day 14: number analyzed (Participants) | 51 | 22
  Day 14 | 1.05 (1.636) | 0.20 (0.646)

7. Secondary Outcome: Rate of Decline in Viral Load
Description: Rate of decline in viral load (Log10 viral particles per milliliter per day [log10 vp/mL/day]) during treatment was measured by qRT-PCR. Viral Load Limit of quantification (LOQ) = 2.18 log10 vp/mL, LOD = 2.05 log10 vp/mL. Results < LOQ and greater than > LOD (target detected) are imputed with 2.12 log10 vp/mL. Results <LOD (target not detected) are imputed with 0 log10 vp/mL.
Time Frame: Up to Day 7
Population: FAS was defined as all randomly assigned participants who received at least 1 dose of study drug and who have a confirmed infection with influenza A.
Measure: Median (95% Confidence Interval); unit: Log10 vp/mL/day
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 63 | 32
Log10 vp/mL/day | -0.35 [-0.39 to -0.30] | -0.42 [-0.49 to -0.35]

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) of Viral Load
Description: Viral load AUC was determined by qRT-PCR assay of nasal swabs. Viral Load LOQ = 2.18 log10 vp/mL, LOD = 2.05 log10 vp/mL. Results <LOQ and >LOD (target detected) are imputed with 2.12 log10 vp/mL. Results <LOD (target not detected) are imputed with 0 log10 vp/mL.
Time Frame: Baseline up to Day 8
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: Days*vp/mL
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 63 | 32
Days*vp/mL | 22.8 [20.4 to 25.1] | 22.1 [19.0 to 25.2]

9. Secondary Outcome: Percentage of Participants With Influenza Complications
Description: Percentage of participants with following Influenza Complications: bacterial pneumonia (culture confirmed where possible), bacterial superinfections, respiratory failure, pulmonary disease (example, asthma, chronic obstructive pulmonary disease [COPD]), cardiovascular and cerebrovascular disease (example, myocardial infarction, congestive heart failure [CHF], arrhythmia, stroke) and all complications were reported.
Time Frame: Up to 28 Days
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 63 | 32
Percentage of participants
  All complications | 7.9 | 15.6
  Bacterial pneumonia | 0 | 0
  Bacterial superinfections | 1.6 | 3.1
  Respiratory failure | 1.6 | 0
  Pulmonary disease | 3.2 | 6.3
  Cardiovascular and Cerebrovascular disease | 1.6 | 0

10. Secondary Outcome: Change From Baseline in Influenza Patient-Reported Outcome Questionnaire (FLU-PRO) Total Score
Description: FLU-PRO assesses 32 influenza symptoms in each of the following body areas (domains): Nose, Throat, Eyes, Chest/Respiratory, Gastrointestinal and Body/Systemic . Participants rate each symptom on a 5-point ordinal scale, with higher scores indicating a more frequent sign or symptom. For 27 of the items, the scale is as follows: 0 ("Not at all"), 1 ("A little bit"), 2 ("Somewhat"), 3 ("Quite a bit"), and 4 ("Very much"). For 5 items, severity is assessed in terms of numerical frequency, that is (i.e), vomiting or diarrhea (0 times, 1 time, 2 times, 3 times, or 4 or more times); with frequency of sneezing, coughing, and coughed up mucus or phlegm evaluated on a scale from 0 ("Never") to 4 ("Always").The FLU-PRO total score is computed as a mean score across all 32 items comprising the instrument. Total scores can range from 0 (symptom free) to 4 (very severe symptoms).
Time Frame: Baseline, Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 31, 32, and 33
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 38 | 32
Units on a scale
  Day 1: number analyzed (Participants) | 20 | 16
  Day 1 | -0.08 (0.247) | -0.11 (0.349)
  Day 2: number analyzed (Participants) | 35 | 20
  Day 2 | -0.48 (0.644) | -0.33 (0.798)
  Day 3: number analyzed (Participants) | 38 | 22
  Day 3 | -0.60 (0.624) | -0.52 (0.641)
  Day 4: number analyzed (Participants) | 35 | 19
  Day 4 | -0.71 (0.702) | -0.56 (0.625)
  Day 5: number analyzed (Participants) | 33 | 17
  Day 5 | -0.76 (0.689) | -0.67 (0.643)
  Day 6: number analyzed (Participants) | 33 | 17
  Day 6 | -0.85 (0.692) | -0.75 (0.659)
  Day 7: number analyzed (Participants) | 33 | 17
  Day 7 | -0.87 (0.738) | -0.69 (0.623)
  Day 8: number analyzed (Participants) | 33 | 18
  Day 8 | -0.89 (0.729) | -0.80 (0.764)
  Day 9: number analyzed (Participants) | 31 | 20
  Day 9 | -0.93 (0.764) | -0.84 (0.732)
  Day 10: number analyzed (Participants) | 32 | 20
  Day 10 | -0.91 (0.723) | -0.81 (0.743)
  Day 11: number analyzed (Participants) | 28 | 18
  Day 11 | -0.87 (0.756) | -0.76 (0.534)
  Day 12: number analyzed (Participants) | 29 | 18
  Day 12 | -0.87 (0.725) | -0.89 (0.695)
  Day 13: number analyzed (Participants) | 28 | 20
  Day 13 | -0.93 (0.702) | -0.94 (0.650)
  Day 14: number analyzed (Participants) | 29 | 19
  Day 14 | -0.85 (0.613) | -0.92 (0.670)
  Day 15: number analyzed (Participants) | 25 | 15
  Day 15 | -0.88 (0.630) | -0.90 (0.724)
  Day 16: number analyzed (Participants) | 23 | 14
  Day 16 | -0.84 (0.588) | -0.90 (0.762)
  Day 17: number analyzed (Participants) | 22 | 15
  Day 17 | -0.98 (0.690) | -0.97 (0.774)
  Day 18: number analyzed (Participants) | 19 | 15
  Day 18 | -1.06 (0.753) | -1.00 (0.868)
  Day 19: number analyzed (Participants) | 21 | 13
  Day 19 | -1.06 (0.749) | -1.05 (0.880)
  Day 20: number analyzed (Participants) | 21 | 15
  Day 20 | -1.03 (0.710) | -1.03 (0.847)
  Day 21: number analyzed (Participants) | 22 | 16
  Day 21 | -1.00 (0.701) | -0.98 (0.849)
  Day 22: number analyzed (Participants) | 18 | 15
  Day 22 | -1.02 (0.789) | -0.92 (0.690)
  Day 23: number analyzed (Participants) | 21 | 14
  Day 23 | -1.11 (0.858) | -0.96 (0.731)
  Day 24: number analyzed (Participants) | 19 | 11
  Day 24 | -0.87 (0.534) | -0.91 (0.580)
  Day 25: number analyzed (Participants) | 17 | 11
  Day 25 | -0.94 (0.659) | -0.85 (0.661)
  Day 26: number analyzed (Participants) | 18 | 11
  Day 26 | -0.86 (0.755) | -0.87 (0.742)
  Day 27: number analyzed (Participants) | 15 | 8
  Day 27 | -1.02 (0.745) | -0.74 (0.734)
  Day 28: number analyzed (Participants) | 12 | 7
  Day 28 | -0.60 (0.505) | -0.82 (0.675)
  Day 29: number analyzed (Participants) | 2 | 2
  Day 29 | -1.13 (0.354) | -1.63 (0.398)
  Day 30: number analyzed (Participants) | 2 | 0
  Day 30 | -0.61 (0.552) |
  Day 31: number analyzed (Participants) | 1 | 0
  Day 31 | -0.75 (NA) — Here, NA indicates that data was not available as standard deviation could not be calculated for a single participant. |
  Day 32: number analyzed (Participants) | 2 | 0
  Day 32 | -0.61 (0.420) |
  Day 33: number analyzed (Participants) | 1 | 0
  Day 33 | -0.94 (NA) — Here, NA indicates that data was not available as standard deviation could not be calculated for a single participant. |

11. Secondary Outcome: Time to Improvement of Vital Signs
Description: Time to improvement of vital signs was defined as the time from first study treatment to when at least 4 of 5 symptoms (temperature, blood oxygen saturation, heart rate, systolic blood pressure, and respiration rate) had recovered, including normalization of temperature and blood oxygen saturation. Resolution criteria for vital signs: for Temperature: oral temperature less than or equal to (<=) 36.5 degree Celsius (C) for elderly and <=37.2 C for adults; for oxygen saturation: greater than or equal to (>=) 92 percent (%) on room air without supplemental oxygen; for respiratory rate: <= 24 per minutes; for heart rate: <= 100 per minutes and for systolic blood pressure: >= 90 millimeters of mercury (mmHg).
Time Frame: Up to 28 Days
Population: FAS was defined as all randomly assigned participants who received at least 1 dose of study drug and who have a confirmed infection with influenza A. Here, N (number of participants analyzed) signifies number of participants evaluable for this OM.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 60 | 28
Hours | 169.92 [46.63 to NA] — Here 'NA' indicates that the upper limit of 95% confidence interval (CI) was not estimable due to less number of events. | 69.90 [35.83 to NA] — Here 'NA' indicates that the upper limit of 95% CI was not estimable due to less number of events.

12. Secondary Outcome: Time to Improvement of Respiratory Status
Description: The time to improvement of respiratory status was defined as the time from first study treatment until the first assessment of a successive series of 3 recording where normalization of blood oxygen saturation and respiration rate occurred at respiration rate <=24 per minutes).
Time Frame: Up to 28 Days
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 60 | 28
Hours | 33.53 [21.33 to 241.92] | 40.57 [22.75 to NA] — Here 'NA' indicates that the upper limit of 95% CI was not estimable due to less number of events.

13. Secondary Outcome: Percentage of Participants With Clinical Outcome Based on Ordinal Scale
Description: The ordinal scale was used to assess participant's clinical outcome. It consists of 6 categories or clinical states that are exhaustive, mutually exclusive, and ordered, where 1- Death, 2- Admitted to intensive care unit (ICU) or mechanically ventilated/ extracorporeal membrane oxygenation (ECMO), 3- Non-ICU plus supplemental oxygen, 4- Non-ICU plus no supplemental oxygen, 5- Not hospitalized, but unable to continue activity, 6- Not hospitalized (NH) and continues activities.
Time Frame: Day 8
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 62 | 31
Percentage of Participants
  Day 8: NH and Continues Activities | 40.3 | 29.0
  Day 8: NH, but Unable to Continue Activity | 27.4 | 45.2
  Day 8: Non-ICU+No Supplemental Oxygen | 14.5 | 6.5
  Day 8: Non-ICU+Supplemental Oxygen | 8.1 | 3.2
  Day 8: Death | 1.6 | 0
  Day 8: Missing | 8.1 | 16.1

14. Secondary Outcome: Number of Participants With the Emergence of Drug Resistance Mutations With Oseltamivir (OST) and Pimodivir
Description: Number of participants with emergence (from baseline) of drug resistance mutations detected by genotype or phenotype were reported.
Time Frame: Up to 28 Days
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 63 | 32
Participants
  Emergence of Pimodivir Mutation | 0 | 0
  Emergence of OST Mutation | 0 | 1

15. Secondary Outcome: Time to Return to Premorbid Functional Status
Description: Time to return to premorbid functional status (time to return usual activities) was defined as time in hours from the first dose of investigational product till the first one of 2 successive cases where the response is 'Yes' on FLU-PRO additional question 7 (Have you returned to your usual activities today?).
Time Frame: Up to Day 33
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 60 | 32
Hours | 142.85 [83.27 to 220.15] | 154.83 [74.97 to 386.52]

16. Secondary Outcome: Time to Hospital Discharge
Description: Time to hospital discharge was calculated from the date of first study drug intake during hospitalization up to date of discharge.
Time Frame: Up to 28 Days
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 63 | 32
Days | 4.00 [3.00 to 5.00] | 4.00 [3.00 to 4.00]

17. Secondary Outcome: Time to Return to Usual Health
Description: Time to return to usual health was defined as the time in hours from the first dose of investigational product till the first one of 2 successive cases where the response is 'Yes' on FLU-PRO additional question 9 (Have you returned to your health today?).
Time Frame: Up to Day 33
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 60 | 32
Hours | 217.05 [122.03 to 291.42] | 338.83 [107.40 to NA] — Here 'NA' indicates that the upper limit of 95% CI was not estimable due to less number of events.

18. Secondary Outcome: Time to Significant Reduction in FLU-PRO Influenza Symptom Severity
Description: Time to significant reduction in influenza symptom severity (mild/none) is time from first dose of investigational drug until first of 2 successive recordings in which total score for each of 2 recordings is lower or equal to 1 and all domain scores is lower or equal to 1. FLU-PRO assesses 32 influenza symptoms in body areas (domains): Nose, throat, eyes, chest, gastrointestinal, body. Participants rate each symptom on 5-point scale, with higher scores indicates more frequent symptom. For 27 of items, scale is as follows: 0 (Not at all), 1 (A little bit), 2 (Somewhat), 3 (Quite a bit), 4 (Very much). For 5 items, severity is assessed in terms of numerical frequency, i.e, vomiting/diarrhea (0 times, 1 time, 2 times, 3 times, or 4 or more times); with frequency of sneezing, coughing and coughed up mucus or phlegm evaluated on scale from 0=Never to 4=Always. FLU-PRO total score is computed as mean score across all 32 items and ranges from 0 (symptom free) to 4 (very severe symptoms).
Time Frame: Up to Day 33
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 60 | 32
Hours | 118.45 [82.33 to 171.93] | 218.72 [94.70 to 275.58]

19. Secondary Outcome: Percentage of Participants With Significant Reduction in FLU-PRO All Influenza Symptoms (Mild or None for All Symptoms)
Description: Percentage of participants with significant reduction in influenza symptom severity was defined as time from first dose of investigational product until first of 2 successive recordings in which FLU-PRO total score for each of 2 recordings <= to 1 and all FLU-PRO domain scores is <=1. FLU-PRO assesses 32 influenza symptoms in body areas (domains): Nose, throat, eyes, chest, gastrointestinal, body. Participants rate each symptom on a 5-point ordinal scale, with higher scores indicates more frequent symptom. For 27 of items, scale is as follows: 0 (Not at all), 1 (A little bit), 2 (Somewhat), 3 (Quite a bit), 4 (Very much). For 5 items, severity is assessed as numerical frequency i.e, vomiting or diarrhea (0-4 or more times); with frequency of sneezing, coughing, coughed up mucus or phlegm evaluated on a scale from 0 (Never)-4 (Always). FLU-PRO total score is computed as a mean score across all 32 items comprising instrument and ranges from 0 (symptom free) to 4 (very severe symptoms).
Time Frame: Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 31, 32 and 33
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
Number analyzed (Participants) | 55 | 30
Percentage of participants
  Day 1: number analyzed (Participants) | 32 | 22
  Day 1 | 9.4 | 18.2
  Day 2: number analyzed (Participants) | 51 | 26
  Day 2 | 37.3 | 34.6
  Day 3 | 36.4 | 26.7
  Day 4: number analyzed (Participants) | 50 | 26
  Day 4 | 42.0 | 38.5
  Day 5: number analyzed (Participants) | 50 | 24
  Day 5 | 54.0 | 37.5
  Day 6: number analyzed (Participants) | 49 | 25
  Day 6 | 59.2 | 40.0
  Day 7: number analyzed (Participants) | 49 | 23
  Day 7 | 55.1 | 34.8
  Day 8: number analyzed (Participants) | 51 | 25
  Day 8 | 62.7 | 32.0
  Day 9: number analyzed (Participants) | 50 | 26
  Day 9 | 76.0 | 38.5
  Day 10: number analyzed (Participants) | 51 | 26
  Day 10 | 76.5 | 53.8
  Day 11: number analyzed (Participants) | 47 | 22
  Day 11 | 70.2 | 59.1
  Day 12: number analyzed (Participants) | 48 | 25
  Day 12 | 77.1 | 72.0
  Day 13: number analyzed (Participants) | 46 | 26
  Day 13 | 76.1 | 69.2
  Day 14: number analyzed (Participants) | 48 | 26
  Day 14 | 77.1 | 65.4
  Day 15: number analyzed (Participants) | 36 | 19
  Day 15 | 63.9 | 57.9
  Day 16: number analyzed (Participants) | 35 | 18
  Day 16 | 71.4 | 66.7
  Day 17: number analyzed (Participants) | 35 | 19
  Day 17 | 74.3 | 63.2
  Day 18: number analyzed (Participants) | 30 | 19
  Day 18 | 70.0 | 57.9
  Day 19: number analyzed (Participants) | 31 | 17
  Day 19 | 77.4 | 58.8
  Day 20: number analyzed (Participants) | 33 | 19
  Day 20 | 81.8 | 63.2
  Day 21: number analyzed (Participants) | 34 | 20
  Day 21 | 79.4 | 60.0
  Day 22: number analyzed (Participants) | 29 | 18
  Day 22 | 86.2 | 61.1
  Day 23: number analyzed (Participants) | 32 | 17
  Day 23 | 78.1 | 70.6
  Day 24: number analyzed (Participants) | 29 | 15
  Day 24 | 86.2 | 66.7
  Day 25: number analyzed (Participants) | 26 | 13
  Day 25 | 92.3 | 69.2
  Day 26: number analyzed (Participants) | 27 | 14
  Day 26 | 81.5 | 57.1
  Day 27: number analyzed (Participants) | 24 | 10
  Day 27 | 83.3 | 50.0
  Day 28: number analyzed (Participants) | 18 | 9
  Day 28 | 77.8 | 44.4
  Day 29: number analyzed (Participants) | 5 | 3
  Day 29 | 80.0 | 66.7
  Day 30: number analyzed (Participants) | 3 | 1
  Day 30 | 100.0 | 0
  Day 31: number analyzed (Participants) | 1 | 0
  Day 31 | 100.0 |
  Day 32: number analyzed (Participants) | 2 | 0
  Day 32 | 100.0 |
  Day 33: number analyzed (Participants) | 1 | 0
  Day 33 | 100 |

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Safety analysis set included all participants who received at least one dose of study drug(s) and were analyzed by drug received.
Arm/Group | Pimodivir 600 mg Plus Oseltamivir 75 mg | Placebo Plus Oseltamivir 75 mg
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/35
Serious Adverse Events (participants affected / at risk) | 11/64 | 4/35
Other Adverse Events (participants affected / at risk) | 45/64 | 24/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimodivir 600 mg Plus Oseltamivir 75 mg (N=64) | Placebo Plus Oseltamivir 75 mg (N=35)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimodivir 600 mg Plus Oseltamivir 75 mg (N=64) | Placebo Plus Oseltamivir 75 mg (N=35)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Amaurosis (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1
Photopsia (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 9 | 5
Oral pain (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 1
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 7 | 3
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT02532283/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02532283/SAP_001.pdf